CLINICAL TRIAL: NCT05812937
Title: The Diagnostic Value of the Intraoperative Intraabdominal Ultrasound for Deep Bowel Endometriosis
Brief Title: Intraoperative Intraabdominal Ultrasound for Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, M.D., University of Palermo
Other Study IDs: INTA-US-ENDO
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Endometriosis; Endometriosis; Bowel; Ultrasound Therapy; Complications
Keywords: Endometriosis; Deep bowel endometriosis; Ultrasound; laparoscopy
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with suspicion of deep bowel endometriosis: Women with suspicion of deep bowel endometriosis undergoing intraoperative ultrasound to assess its diagnostic value for endometriosis patients as well as the predictive potential of changing the therapeutic strategy during the surgery based on the ultrasound findings.
  Interventions: Procedure: Intraabdominal ultrasound

INTERVENTIONS:
Procedure: Intraabdominal ultrasound — To assess the diagnostic value of the intraoperative intrabaabdominal ultrasound (IIUS) for endometriosis patients as well as the predictive potential of changing the therapeutic strategy during the surgery based on the ultrasound findings.
  Other Names: Laparoscopic visualization; Laparoscopic palpation; Direct palpation in case of a conventional segmental bowel resection with specimen extraction per minilaparotomy.

SUMMARY:
The diagnosis of bowel endometriosis lesions is in most cases a combination of anamnesis, clinical exam, transvaginal ultrasound (and/or MRI and/or endorectal sonography) and laparoscopy.

Both the transvaginal ultrasound as well as the MRI have showed a great accuracy with very good sensititivity and specificity regarding the imaging diagnosis of bowel endometriosis.

The conventional laparoscopy contributes to the diagnosis of bowel endometriosis by visualizing the nodules and palpating the deep endometriosis nodule using the instruments, therefor offering the surgeon a haptic feedback by grasping, pushing and rolling the bowel wall and the nodules. Horace Roman and Dan Martin showed that 25% of patients undergoing a conventional laparoscopic segmental bowel resection with a minilaparotomy hat palpable non-visualized endometriosis nodules. These nodules could be directly palpated with the hands because the bowel was exteriorized through the minilaparotomy. The direct palpation of the bowel offers of course a superior haptic feedback compared to the haptic feedback offered by the laparoscopic palpation using the instruments. However this was a direct palpation of only the oral part of the bowel. The aboral part of the bowel caudal to the staple line could not be evaluated by direct palpation. New surgical techniques for the segmental bowel resection with transvaginal/transanal NOSE(natural orifice specimen extraction) have been described in the last years. The novel techniques avoid the minilaparotomy and assure a 100% minimal invasive approach offering better esthetic outcomes.

However in such cases a direct palpation of the bowel wall using the hands in order to identify non- visualizable nodules is not possible as the bowel remains the whole time of the procedure inside of the abdomen. On the other side the robotic-assisted laparoscopy doesn't offer the surgeon a haptic feedback at all. In these cases the surgeon has to rely on the visual aspects of the lesions and therefor "touch" the lesions with his eyes - the visual information should replace the haptic feedback. So in the case of a robotic assisted laparoscopic segemental bowel resection with a NOSE it is not possible to palpate the bowel at all - neither with instruments, not with the hands. Other surgical techniques used to excise smaller colorectal nodules are the rectal shaving and the full thickness excision (disc excision) using a circular stapler. In these situations the surgeon has to rely exclusively on the visual information as well on the haptic feedback given by the conventional laparoscopic instruments. In more than 30% of the cases of full thickness rectal resection the resection the margins are infiltrated by the endometriosis nodules. All the above mentioned situations raise the question of the radicallity in terms of healthy resection margins and of multifocal lesions that cannot be visualized and/or palpated. In this study we are evaluating the diagnostic value of the intraoperative intraabdominal ultrasound for deep infiltrating colorectal endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with suspicion of endometriosis who undergo surgery.

Exclusion Criteria:

* Patients under 18 years old;
* Patients who didn't sign the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women affected by deep bowel endometriosis.
Study Population: Women affected by deep bowel endometriosis undergoing intraabdominal ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of IIUS compared to TVS regarding the colorectal endometriosis | At the moment of the surgery
  Compare the dimmensions of preop. TVS-diagnosed nodules with the intraop. IUS dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Alin Constantin, M.D., Principal Investigator — Albertinen Hospital Hamburg; Antonio Simone Laganà, M.D. Ph.D., Study Director — University of Palermo; Andrea Etrusco, M.D., Study Chair — University of Palermo; Vito Chiantera, M.D. Ph.D., Study Chair — University of Palermo
Locations (1):
- Albertinen Hospital, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No